CLINICAL TRIAL: NCT06675006
Title: Comparative Analysis of Cryotherapy Combined With Bowen Therapy Versus Medical Massage for Managing Acute Ankle Sprain
Brief Title: Comparing Bowen Therapy With Ice to Medical Massage for Acute Ankle Sprain
Acronym: ICE-BOW
Status: Completed | Type: Observational
Sponsor: Rehabilitation Centre Zivot (Other)
Responsible Party: Principal Investigator, Darko Bilic, Director, Rehabilitation Centre Zivot
Other Study IDs: B2024
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Ankle Sprains
Keywords: Bowen therapy; Cryotherapy
MeSH Terms: conditions — Ankle Injuries | interventions — Cryotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bowen Therapy with Cryotherapy Group: This group consists of participants receiving Bowen therapy combined with cryotherapy for the treatment acute ankle sprain. Each session includes a 30-minute Bowen therapy treatment, focusing on gentle, non-invasive movements designed to stimulate the body's healing processes. Cryotherapy involves the application of ice to the affected area to reduce inflammation and pain. Participants in this group will undergo three treatment sessions on days 1, 8, and 15 of the study, with assessments of pain intensity and functional capacity conducted before and after the intervention.
- Medical Massage and Cryotherapy Group: This group consists of participants who receive traditional medical massage for the treatment of acute ankle sprain. Interventions are conducted over three sessions, occurring on days 1, 8, and 15, with each session lasting 30 minutes. The medical massage aims to alleviate pain, improve muscle relaxation, and enhance overall functionality in daily activities. Participants' pain levels and functional capacity are assessed using the VAS pain scale and Roland-Morris questionnaire at both the beginning and end of the study period.
  Interventions: Combination Product: Medical Massage

INTERVENTIONS:
Combination Product: Medical Massage — This intervention refers to the application of therapeutic massage techniques aimed at alleviating pain and enhancing muscle relaxation in patients with nonspecific low back pain. The treatment focuses on manipulating soft tissues, including muscles, tendons, and fascia, to improve circulation, reduce muscle tension, and promote overall wellness. Medical massage is tailored to each patient's specific needs and can incorporate various techniques, including Swedish massage, Bowen Therapy, a gentle and non-invasive manual therapy, utilizes precise movements on specific points of the body to promote healing and restore balance. The therapist applies light pressure with the fingers, allowing the body to respond and relax. This technique aims to stimulate the body's innate healing mechanisms, encouraging improvements in pain levels and functional capacity. Sessions are typically structured to allow for periods of rest, giving the body time to process the treatment and enhancing its effects.
  Other Names: Bowen therapy; Cryotherapy
  Groups: Medical Massage and Cryotherapy Group

SUMMARY:
Foot pain is particularly prevalent among older adults, affecting approximately 20% to 37% of men and women aged 45 years and older living in the community. Ankle pain is somewhat less common. This study evaluates the combined impact of cryotherapy (ice application) with Bowen therapy versus traditional medical massage in alleviating symptoms. A total of 41 patients, aged 32-75 years participated and were divided into two treatment groups: one receiving medical massage and ice, and the other Bowen therapy and ice, with three sessions over 15 days. Pain and functionality were measured using the VAS pain scale and Roland-Morris questionnaire. Findings revealed improvements in both groups, with the Bowen therapy group achieving greater pain reduction and functional improvement, suggesting potential advantages of Bowen therapy combined with cryotherapy for managing symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 32 to 75 years.
* Diagnosed with ankle sprain by a qualified healthcare professional (physiatrist or orthopedist).
* Able to provide informed consent.
* Willing to comply with the study protocol and attend all scheduled therapy sessions.

Exclusion Criteria:

* Presence of serious spinal pathologies (e.g., cancer, osteoporosis, trauma, or fracture).
* History of significant neurological disorders or conditions affecting mobility.
* Pregnancy or breastfeeding.
* Previous surgical interventions on the spine or significant other surgeries within the last six months.
* Current use of medications that affect pain perception (e.g., opioids).
* Participation in other therapeutic interventions for low back pain during the study period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of 40 adult participants aged between 32 and 75 years, with a mean age of 52.1 years (SD ± 10.6). Participants are randomly assigned to two groups: one receiving Bowen therapy and the other receiving medical massage, allowing for a comparative analysis of the efficacy of each intervention. All participants provided informed consent prior to enrollment in the study and are expected to attend all scheduled therapy sessions and follow-up assessments.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Pain Intensity Reduction | 15 days
  Pain intensity will be assessed using the Visual Analog Scale (VAS), which allows participants to rate their pain on a scale from 0 (no pain) to 10 (worst possible pain). This measure will be taken at baseline (Day 1) and at the end of the intervention period (Day 15) to evaluate the effectiveness of the interventions in reducing pain levels.

SECONDARY OUTCOMES:
Functional Improvement | 15 days
  Functional status will be evaluated using the Roland-Morris Disability Questionnaire, which assesses the impact of ankle sprain on daily activities. Participants will complete this questionnaire at the start of the study and upon completion of the intervention to determine changes in functional ability and quality of life.

OTHER OUTCOMES:
Patient Satisfaction | 15 days
  Participants will provide feedback regarding their satisfaction with the treatment received through a brief questionnaire administered at the end of the study. This will include questions related to their overall experience with the therapy, perceived effectiveness, and likelihood of recommending the treatment to others.

CONTACTS AND LOCATIONS:
Locations (1):
- Rehabilitation Centre Život, Mostar, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Amjad F, Khalid A. Comparative effects of Bowen therapy and tennis ball technique on pain and functional disability in patients with thoracic myofascial pain syndrome. J Orthop Surg Res. 2023 Nov 24;18(1):895. doi: 10.1186/s13018-023-04379-z. PMID 37996838
- [Background] Marr M, Baker J, Lambon N, Perry J. The effects of the Bowen technique on hamstring flexibility over time: a randomised controlled trial. J Bodyw Mov Ther. 2011 Jul;15(3):281-90. doi: 10.1016/j.jbmt.2010.07.008. Epub 2010 Sep 15. PMID 21665103
- [Background] Sivakumar P, Dhinakaran S, Sudharshini. Bowen Therapy: An Overview. Pon J Nurs. 2022;15(1):16-18.
- [Background] Tikhile P, Patil DS. Unveiling the Efficacy of Physiotherapy Strategies in Alleviating Low Back Pain: A Comprehensive Review of Interventions and Outcomes. Cureus. 2024 Mar 12;16(3):e56013. doi: 10.7759/cureus.56013. eCollection 2024 Mar. PMID 38606230
- [Background] Shokri P, Zahmatyar M, Falah Tafti M, Fathy M, Rezaei Tolzali M, Ghaffari Jolfayi A, Nejadghaderi SA, Sullman MJM, Kolahi AA, Safiri S. Non-spinal low back pain: Global epidemiology, trends, and risk factors. Health Sci Rep. 2023 Sep 4;6(9):e1533. doi: 10.1002/hsr2.1533. eCollection 2023 Sep. PMID 37674621